CLINICAL TRIAL: NCT01588184
Title: A Single Arm, Open Label Multicentre Extension Study of Bevacizumab in Patients With Solid Tumours on Study Treatment With Bevacizumab, at the End of A F. Hoffmann-La Roche and/or Genentech Sponsored Study
Brief Title: An Extension Study to Provide Continued Bevacizumab Therapy to Participants With Solid Tumors Who Were Previously Enrolled in a Roche/Genentech Sponsored Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO25757; 2011-002009-31 (EudraCT Number)
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: All participants were assigned the same treatment. The Number of Arms represent the reporting groups of all subjects according to disease.

ARMS (6):
- Breast Cancer (Experimental): Participants will receive bevacizumab until progression of disease or unacceptable toxicity, withdrawal of consent or death whichever occurs first.
  Interventions: Drug: Bevacizumab
- Ovarian Cancer or Peritoneal Carcinoma (Experimental): Participants will receive bevacizumab until progression of disease or unacceptable toxicity, withdrawal of consent or death whichever occurs first.
  Interventions: Drug: Bevacizumab
- Renal Cell Carcinoma (Experimental): Participants will receive bevacizumab until progression of disease or unacceptable toxicity, withdrawal of consent or death whichever occurs first.
  Interventions: Drug: Bevacizumab
- Colorectal Cancer (Experimental): Participants will receive bevacizumab until progression of disease or unacceptable toxicity, withdrawal of consent or death whichever occurs first.
  Interventions: Drug: Bevacizumab
- Non-Squamous, Non-Small Cell Lung Cancer (Experimental): Participants will receive bevacizumab until progression of disease or unacceptable toxicity, withdrawal of consent or death whichever occurs first.
  Interventions: Drug: Bevacizumab
- Glioblastoma Multiforme (Experimental): Participants will receive bevacizumab until progression of disease or unacceptable toxicity, withdrawal of consent or death whichever occurs first.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered at 7.5 or 15 milligrams per kilogram (mg/kg) intravenously every 3 weeks (Q3W), or 5 or 10 mg/kg intravenously every 2 weeks (Q2W).
  Other Names: Avastin

SUMMARY:
This single-arm, open-label, multicenter extension study will provide continued bevacizumab therapy to participants with solid tumors who were previously enrolled in a Roche/Genentech sponsored study and who derived benefit from the bevacizumab therapy. Participants will receive the same dose and regimen of bevacizumab as used in the previous parent trial and continue this treatment until progression of disease or unacceptable toxicity, withdrawal of consent or death whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Participant is treated with bevacizumab at the end of the Roche/Genentech sponsored parent trial and continues to have benefit as judged by the investigator
* Eligible for continuation of bevacizumab treatment at the end of a parent trial, according to parent trial protocol
* Able to comply with this extension study protocol (MO25757)

Exclusion Criteria:

* Evidence of disease progression assessed according to parent trial protocol during the screening phase for this extension study
* Evidence of any adverse event potentially attributable to bevacizumab, for which the local label recommends permanent discontinuation
* A treatment interruption with bevacizumab of more than 42 days since the last administration of bevacizumab in the parent trial
* Evidence of any other disease that would put the participant at high risk for treatment-related complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2012-07-13 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (73):
- A.Ö. LKH; Abt. für Lungenkrankheiten, Steyr, Austria
- Brazil (7):
  - Hospital Araujo Jorge; Departamento de Ginecologia E Mama, Goiânia, Goiás
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Perola Byington, São Paulo, São Paulo
  - Hospital A. C. Camargo; Oncologia, São Paulo, São Paulo
  - Hospital Sao Jose, São Paulo, São Paulo
- MBAL Serdika EOOD, Sofia, Bulgaria
- University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario, Canada
- Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc, Czechia
- North Estonia Medical Centre Foundation; Oncology Center, Tallinn, Estonia
- France (7):
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Centre Leonard De Vinci;Chimiotherapie, Dechy
  - Centre Georges François Leclerc; Service Pharmacie, Bp 77980, Dijon
  - Hopital Roger Salengro; Service de Neurologie, Lille
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Centre Paul Strauss; Oncologie Medicale, Strasbourg
  - Hopital Larrey; Pneumologie, Toulouse
- Germany (2):
  - Klinikum Joh.Wolfg.Goethe-UNI Senckenbergisches Institut für Neuroonkologie, Frankfurt am Main
  - LungenClinic Großhansdorf GmbH, Großhansdorf
- Orszagos Onkologiai Intezet; Nogyogyaszati Osztaly, Budapest, Hungary
- Italy (13):
  - Ospedale Antonio Perrino; Oncologia Medica, Brindisi, Apulia
  - A.O. Universitaria Federico II Di Napoli; Oncologia Ed Endocrinologia Clinica, Napoli, Campania
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi; Unità Operativa Oncologia Medica, Bologna, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini; U.O.C. Pneumologia Ad Indirizzo Oncologico 1, Rome, Lazio
  - Fondazione IRCCS Istituto Neurologico C. Besta; Neuro-oncologia Sperimentale e Terapia Genica, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Oncologia Medica, Milan, Lombardy
  - ASST DI MONZA; Oncologia Medica, Monza, Lombardy
  - ASST LARIANA; Oncologia, S. Fermo Della Battaglia (CO), Lombardy
  - Azienda Ospedaliera Le Molintte di Torino; Dipartimento Di Neurologia - Oncologia, Turin, Piedmont
  - Centro Catanese Di Oncologia; Oncologia Medica, Catania, Sicily
  - Ospedale Nuovo Della Versilia; Divisione Di Oncologia Medica, Lido di Camaiore, Tuscany
  - A.O. Universitaria Pisana-Ospedale Cisanello; Dipartimento Cardio Toracico-Pneumologia Ii, Pisa, Tuscany
  - Ospedale Misericordia E Dolce; Oncologia Medica, Prato, Tuscany
- Mexico (3):
  - Instituto Nacional de Cancerologia; Oncology, Distrito Federal
  - Fundación Rodolfo Padilla Padilla, A.C.; Oncology, León
  - Oaxaca Site Management Organization, Oaxaca City
- Netherlands (2):
  - Radboud Ziekenhuis; Urologie, 659, Nijmegen
  - Leyenburg Hospital; Pulmonology, The Hague
- Romania (2):
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - Euroclinic Center of Oncology SRL, Iași
- Russia (8):
  - Altai Region Oncology Dispensory; Oncology, Barnaul
  - Regional Oncology Hospital; Oncology, Irkutsk
  - Blokhin Cancer Research Center; Combined Treatment, Moscow
  - Russian Research Center of Roentgenoradiology; Dept of Chemotherapy, Moscow
  - P.A. Gertsen Cancer Research Inst. ; Chemotherapy Dept, Moscow
  - City Clinical Oncology Hospital, Moscow
  - Medical Radiological Scientific Center; Department of Radiotherapy of Gynaecological Disease, Obninsk, Kaluzhskaya Region
  - Bashkirian Republican Clinical Oncology Dispensary, Ufa
- Vychodoslovensky onkologicky ustav, Košice, Slovakia
- Wits Donald Gordon Clinical Trial Centre; Medical Oncology, Parktown, Johannesburg, South Africa
- South Korea (3):
  - National Cancer Center; Medical Oncology, Gyeonggi-do
  - Severance Hospital; Internal Medicine, Seoul
  - Asan Medical Center, Uni Ulsan Collegemedicine; Dept.Internal Medicine / Divisionhematology/Oncology, Seoul
- Spain (11):
  - Hospital de Basurto; Servicio de Oncologia, Bilbao, Vizcaya
  - Hospital de Cruces; Servicio de Oncologia, Bilbao, Vizcaya
  - Complejo Hospitalario Universitario A Coruña (CHUAC, Materno Infantil), Oncología, A Coruña
  - Complejo Asistencial Universitario De Burgos; Servicio de Oncologia, Burgos
  - Hospital Reina Sofia; Medical Oncology, Córdoba
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Hospital Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Regional Universitario Carlos Haya; Servicio de Oncologia, Málaga
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
- Sweden (3):
  - Mälarsjukhuset, Eskilstuna, Kvinnokliniken, Eskilstuna
  - Universitetssjukhuset Örebro, Onkologiska kliniken, Örebro
  - Norrlands universitetssjukhus; Onkologkliniken, Umeå
- Adana City Hospital, Medical Oncology, Adana, Turkey (Türkiye)
- United Kingdom (3):
  - Addenbrooke'S Hospital; Dept of Neurosurgery, Cambridge
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester
  - North Wales Cancer Treatment Centre, Glan Clwyd Hospital, Rhyl

REFERENCES:
- [Derived] Oza AM, Dubois F, Hegg R, Hernandez CA, Finocchiaro G, Ghiringhelli F, Zamagni C, Nick S, Irahara N, Perretti T, Colombo N. A Long-Term Extension Study of Bevacizumab in Patients With Solid Tumors. Oncologist. 2021 Dec;26(12):e2254-e2264. doi: 10.1002/onco.13971. Epub 2021 Oct 4. PMID 34498344

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants enrolled over the planned recruitment period was open. 95 participants actually enrolled in this study.
Period: Overall Study
Arm/Group | Breast Cancer | Ovarian Cancer or Peritoneal Carcinoma | Colorectal Cancer | Renal Cell Carcinoma | Non-Squamous, Non-Small Cell Lung Cancer | Glioblastoma Multiforme
Started | 11 | 41 | 7 | 6 | 16 | 14
Completed | 8 | 28 | 5 | 3 | 14 | 10
Not Completed | 3 | 13 | 2 | 3 | 2 | 4
Not completed — Death | 1 | 0 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 4 | 0 | 1 | 0 | 0
Not completed — Bevacizumab treatment provision changed | 0 | 6 | 2 | 0 | 1 | 3
Not completed — multiple reasons | 0 | 3 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Breast Cancer | Ovarian Cancer or Peritoneal Carcinoma | Colorectal Cancer | Renal Cell Carcinoma | Non-Squamous, Non-Small Cell Lung Cancer | Glioblastoma Multiforme | Total
Number analyzed (Participants) | 11 | 41 | 7 | 6 | 16 | 14 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (7.3) | 56.7 (11.2) | 66.7 (13.9) | 63.5 (9.8) | 58.5 (10.5) | 49.5 (10.9) | 56.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 41 | 3 | 2 | 6 | 4 | 67
  Male | 0 | 0 | 4 | 4 | 10 | 10 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 11 | 41 | 7 | 6 | 16 | 14 | 95

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.
Time Frame: Baseline up to approximately 81 months
Measure: Number; unit: percentage of participants
Arm/Group | Breast Cancer | Ovarian Cancer or Peritoneal Carcinoma | Colorectal Cancer | Renal Cell Carcinoma | Non-Squamous, Non-Small Cell Lung Cancer | Glioblastoma Multiforme
Number analyzed (Participants) | 11 | 41 | 7 | 6 | 16 | 14
percentage of participants | 90.9 | 78.0 | 71.4 | 100.0 | 75.0 | 83.2

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as the time from first dose of Bevacizumab in this extension trial (E-trial) to the time of first documented disease progression or death due to any cause, whichever occurs first.
Time Frame: Baseline up to approximately 81 months
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Breast Cancer | Ovarian Cancer or Peritoneal Carcinoma | Colorectal Cancer | Renal Cell Carcinoma | Non-Squamous, Non-Small Cell Lung Cancer | Glioblastoma Multiforme
Number analyzed (Participants) | 11 | 41 | 7 | 6 | 16 | 14
months | 35.31 (23.809) | 24.39 (19.759) | 17.98 (24.202) | 9.31 (12.046) | 17.14 (14.152) | 11.31 (10.301)

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival time is defined as the time from first dose of Bevacizumab in the E-trial to death from any cause.
Time Frame: Baseline up to approximately 81 months
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Breast Cancer | Ovarian Cancer or Peritoneal Carcinoma | Colorectal Cancer | Renal Cell Carcinoma | Non-Squamous, Non-Small Cell Lung Cancer | Glioblastoma Multiforme
Number analyzed (Participants) | 11 | 41 | 7 | 6 | 16 | 14
months | 38.82 (24.159) | 27.35 (20.020) | 20.30 (23.761) | 11.98 (10.950) | 18.31 (14.962) | 12.99 (10.795)

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 81 months
Arm/Group | Breast Cancer | Ovarian Cancer or Peritoneal Carcinoma | Colorectal Cancer | Renal Cell Carcinoma | Non-Squamous, Non-Small Cell Lung Cancer | Glioblastoma Multiforme
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/41 | 0/7 | 1/6 | 1/16 | 1/14
Serious Adverse Events (participants affected / at risk) | 2/11 | 2/41 | 2/7 | 3/6 | 5/16 | 3/14
Other Adverse Events (participants affected / at risk) | 10/11 | 31/41 | 5/7 | 6/6 | 12/16 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Breast Cancer (N=11) | Ovarian Cancer or Peritoneal Carcinoma (N=41) | Colorectal Cancer (N=7) | Renal Cell Carcinoma (N=6) | Non-Squamous, Non-Small Cell Lung Cancer (N=16) | Glioblastoma Multiforme (N=14)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COMPLICATED APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MENINGITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
JAW FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Breast Cancer (N=11) | Ovarian Cancer or Peritoneal Carcinoma (N=41) | Colorectal Cancer (N=7) | Renal Cell Carcinoma (N=6) | Non-Squamous, Non-Small Cell Lung Cancer (N=16) | Glioblastoma Multiforme (N=14)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 5 (20) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (7) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 3 (9) | 1 (12) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHILIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 3 (10) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LACRIMATION INCREASED (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERIORBITAL DISORDER (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
XEROPHTHALMIA (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (21) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEILITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 7 (19) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 5 (8) | 0 (0) | 0 (0) | 3 (7) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PEPTIC ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 4 (5) | 3 (5) | 0 (0) | 0 (0) | 3 (5) | 5 (6)
CHEST PAIN (General disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 4 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 4 (7) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
CONTRAST MEDIA ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEASONAL ALLERGY (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERIURIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BREAST DISCHARGE INFECTED (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LACRIMAL GLAND ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAIL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PERIODONTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RHINITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 9 (26) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
AMYLASE INCREASED (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (3) | 2 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 5 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
EJECTION FRACTION DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIPASE INCREASED (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 (1) | 4 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 4 (7) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
APHONIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COMPLEX REGIONAL PAIN SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSTONIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FACIAL NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 3 (5) | 4 (6) | 1 (1) | 0 (0) | 1 (1) | 6 (7)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MOVEMENT DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUROTOXICITY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
IRRITABILITY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 6 (55) | 20 (100) | 2 (5) | 1 (1) | 8 (26) | 5 (15)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CYSTOCELE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN SWELLING (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH EXTRACTION (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EMBOLISM VENOUS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 2 (3) | 7 (25) | 0 (0) | 2 (5) | 1 (1) | 0 (0)
LYMPHOEDEMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT01588184/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT01588184/SAP_001.pdf